CLINICAL TRIAL: NCT02221843
Title: An Observational Single Center Pilot Study Using a Wearable UV Sensor (Sunbit) Measuring UV Exposure of Patients at High Risk for Skin Cancer - SUNBIT Study
Brief Title: Sunbit UV Measuring Device to Track Sun Behavior
Status: Terminated | Type: Observational
Why Stopped: Company dissolved, no study devices available anymore
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK2013-0283_Sunbit
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Immunosuppression; Skin Neoplasms
Keywords: sun behavior; immunosuppression; skin neoplasms; sunbit; uv sensor; uv dosimeter; solar radiation; uv exposition; uv index
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sunbit is a new wearable UV dosimeter to measure solar radiation in real time. The purpose of this study is to track sun behavior of patients at high risk for skin cancer, to investigate the feasibility of this prototype in daily life and to investigate the technical accuracy of the Sunbit.

DETAILED DESCRIPTION:
A total of 20 patients will be included to wear the Sunbit system during the time of 4 weeks. After this 4 weeks Sunbit will be recollected and data in the form of UV Indices will be extracted and analyzed.

Patients will be recruited in the Department of Dermatology of the University Hospital Zürich. The target population comprises patients with a high risk of melanoma and non-melanoma skin cancer, thus especially patients with an immunosuppressive therapy due to organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* History of skin cancer (melanoma or NMSC) or patients with high risk of skin cancer (e.g. immunosuppressive therapy)
* Oral and written informed consent

Exclusion Criteria:

* Any medical condition that renders the patient bedridden for the duration of 2 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Dermatology of the University Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
number of days wearing the device | after 4 weeks wearing the device
  patient compliance

SECONDARY OUTCOMES:
difference between measured UV Indices and reference values | after 4 weeks wearing the device
  technical accuracy of the device

OTHER OUTCOMES:
difference between the individual UV Indices | after 4 weeks wearing the device
  sun behavior

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, Prof. MD, Principal Investigator — Department of Dermatology of the University Hospital Zurich
Locations (1):
- Department of Dermatology of the University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
none intended

REFERENCES:
- See also: Fahrni, T. Sundroid (renamed Sunbit): Solar Radiation Awareness with Smartphones. 2011 — http://www.tik.ee.ethz.ch/file/0be29fd9c90eabb3b0772f37535ef29b/ubicomp11_237.pdf.